CLINICAL TRIAL: NCT00141960
Title: YM1170 Phase 2/3 Study: A Double Blind, Placebo Controlled, Group-comparison Study in Patients With Non-erosive Gastroesophageal Reflux Disease
Brief Title: Famotidine in Subjects With Non-erosive Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1170-CL-004
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2010-06

CONDITIONS: Gastroesophageal Reflux
Keywords: Treatment efficacy; Treatment effectiveness; Gastrointestinal Diseases; Reflux, Gastroesophageal; GERD
MeSH Terms: conditions — Gastroesophageal Reflux; Gastrointestinal Diseases | interventions — Famotidine

INTERVENTIONS:
Drug: Famotidine

SUMMARY:
Gastroesophageal reflux disease (GERD) considered to be associated with mucosal damages in the esophagus and heartburn, which may sometimes interfere with daily activities due likely to reflux of acid gastric contents. While most of the patients given the diagnosis of GERD do not exhibit endoscopically obvious impairment in esophageal mucous membrane, they have subjective symptoms of non-erosive GERD including heartburn. But no drug has been launched in Japan, which targets non-erosive GERD. This study will examine the efficacy and safety of famotidine in subjects with non-erosive GERD.

ELIGIBILITY:
Inclusion Criteria:

* Patients have heartburn with non-erosive gastroesophageal reflux disease.

Exclusion Criteria:

* Patients have diseases which interfere with evaluation of the efficacy and safety in this study.
* Patients are receiving and/or have received prior to the enrollment the treatment which interfere with evaluation of the efficacy and safety in this study.
* Patients have severe cardiovascular, hepatic, renal and hematological disorders.
* Patients are allergic to or have a history of drug allergy to H2RA.
* Patients have or have a history of malignant tumors.
* Patients are pregnant or a lactating mother.
* Patients have participated in other clinical studies less than 12 weeks prior to submitting the informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2005-09

PRIMARY OUTCOMES:
Rate of days with no heart burn in the treatment period

SECONDARY OUTCOMES:
Disappearance of heart burn
Severity of heart burn
Frequency of heart burn
Patient's final global improvement rating
Other symptoms (e.g.,reflux sensation of gastric fluid, discomfort of pharynges)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Chair — Clinical Development III, Astellas Pharm. Inc.
Locations (7):
- Japan (7):
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region
  - Tokai Region

REFERENCES:
- [Background] Hongo M, Kinoshita Y, Haruma K. A randomized, double-blind, placebo-controlled clinical study of the histamine H2-receptor antagonist famotidine in Japanese patients with nonerosive reflux disease. J Gastroenterol. 2008;43(6):448-56. doi: 10.1007/s00535-008-2186-5. Epub 2008 Jul 4. PMID 18600389